CLINICAL TRIAL: NCT03583606
Title: A Systems Biology Phase 1 Evaluation of the Safety, Reactogenicity, and Immunogenicity of Chimpanzee Adenovirus Type 3- Vectored Zaire Ebolavirus (ChAd3-EBO-Z) and Modified Vaccinia Ankara- Vectored Multivalent Filovirus (MVA-BN(R)-Filo) Vaccine Candidates
Brief Title: A Trial to Evaluate the Safety and Systems Biology Response of Ebolavirus Zaire Vaccine (ChAd3-EBO-Z)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 14-0092
Record Dates: First submitted 2018-06-28; First posted 2018-07-11 (Actual); Results first posted 2021-06-02 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2020-07-15

CONDITIONS: Ebola Disease; Immunisation
Keywords: Adenovirus vector; Ebola Virus; Immunogenicity; Non-Human Primates Vaccination/Challenge Studies; Phase 1; Reactogenicity; Safety; Zaire ebolavirus vaccine
MeSH Terms: conditions — Hemorrhagic Fever, Ebola

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- ChAd3-EBO-Z + ChAd3-EBO-Z (Experimental): ChAd3-EBO-Z (2 x 10^11 virus particles (vp)) intramuscularly into the deltoid on Day 1 and ChAd3-EBO-Z (2 x 10^11 vp) intramuscularly into the opposite arm on Day 8, n = 20
  Interventions: Biological: ChAd3-EBO-Z
- ChAd3-EBO-Z + Placebo (Experimental): ChAd3-EBO-Z (2 x 10^11 virus particles (vp)) intramuscularly into the deltoid on Day 1 and placebo intramuscularly into the opposite arm on Day 8, n = 20
  Interventions: Biological: ChAd3-EBO-Z; Other: Placebo
- ChAd3-EBO-Z + MVA- BN-Filo (Experimental): ChAd3-EBO-Z (2 x 10^11 virus particles (vp)) intramuscularly into the deltoid on Day 1 and MVA-BN-Filo (1 x 10^8 Infectious Units (IU)) intramuscularly into the opposite arm on Day 8, n = 20
  Interventions: Biological: ChAd3-EBO-Z; Biological: MVA Multi-Filo Ebola Vaccine

INTERVENTIONS:
Biological: ChAd3-EBO-Z — Zaire ebolavirus vaccine administered by an IM injection into the deltoid as a single dose of 2 x 10^11 virus particles (vp)).
Biological: MVA Multi-Filo Ebola Vaccine — A booster vaccination of replication defective MVA-BN-Filo administered by an IM injection into the deltoid as a single dose of 1 x 10^8 Infectious Units (IU).
  Arms: ChAd3-EBO-Z + MVA- BN-Filo
Other: Placebo — 0.5 mL normal saline administered via IM injection into the deltoid.
  Arms: ChAd3-EBO-Z + Placebo

SUMMARY:
This initial, proof of concept study will focus on identifying significant differences in response to the Ebolavirus Zaire vaccine (ChAd3-EBO-Z) when administered with placebo, MVA-BN(R)-Filo, or ChAd3-EBO-Z boosters after 8 days. All 60 participants will receive the ChAd3-EBO-Z vaccine and then randomized into each booster group (20 receiving each type of booster). Subjects will be followed-up for 6 months to monitor for safety outcomes and efficacy measures. There is no formal hypothesis for this study. The primary objective of this study is to assess the safety and reactogenicity of study products by study group when administered IM to healthy adults.

DETAILED DESCRIPTION:
This is a Phase 1, randomized, double-blind trial of 60 evaluable males and non-pregnant females, 18-45 years old, inclusive, who are in good health, meet all eligibility criteria, and do not meet any exclusion criteria. This trial is designed to assess the safety, reactogenicity and immunogenicity of an Ebolavirus Zaire (ChAd3-EBO-Z) vaccine for the prevention of Ebola. ChAd3-EBO-Z will be administered intramuscularly into the deltoid of all participants on Day 1. On Day 8, subjects will receive either placebo, ChAd3-EBO-Z , or MVA- BN(R)-Filo boosters, administered intramuscularly into the deltoid of the arm opposite their first vaccination, based on study group. There will be 20 subjects in each group. Subjects will be monitored for 6 months after vaccination to assess safety and efficacy for ChA3d-EBO-Z with homologous and heterologous boosting. Differences between the homologous and heterologous arm represent potential points for further, more in depth assessment to determine if there is a correlation with efficacy. Long term goals include comparing results from this study with results from naturally infected individuals as well as non-human primate (NHP) vaccination/challenge studies. There is no formal hypothesis for this study. The primary objective of this study is to assess the safety and reactogenicity of study products by study group when administered IM to healthy adults. The secondary study objective is to assess the antibody response to Zaire ebolavirus (EBOV) glycoprotein (GP) by study group.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent before initiation of any study procedures.
2. Are able to understand and comply with planned study procedures and be available for all study visits/phone calls.
3. Males or non-pregnant females ages 18-45, inclusive.
4. Subject must have a body mass index (BMI) > / = 18.5 and < 35 kg/m^2.
5. Are in good health.

   * As determined by medical history and physical examination to evaluate acute or currently ongoing chronic medical diagnoses or conditions, defined as those that have been present for at least 90 days which would affect the assessment of the safety of subjects or the immunogenicity of study vaccinations. Chronic medical diagnoses or conditions should be stable for the last 60 days (no hospitalizations, ER or urgent care for condition and no adverse symptoms that need medical intervention such as medication change/supplemental oxygen). This includes no change in chronic prescription medication, dose, or frequency as a result of deterioration of the chronic medical diagnosis or condition in the 60 days prior to enrollment. Any prescription change that is due to change of health care provider, insurance company, etc., or that is done for financial reasons, as long as in the same class of medication, will not be considered a deviation of this inclusion criterion. Any change in prescription medication due to improvement of a disease outcome, as determined by the site principal investigator or appropriate sub-investigator, will not be considered a deviation of this inclusion criterion. Subjects may be on chronic or as needed (prn) medications if, in the opinion of the site principal investigator or appropriate sub-investigator, they pose no additional risk to subject safety or assessment of reactogenicity and immunogenicity and do not indicate a worsening of medical diagnosis or condition. Similarly, medication changes subsequent to enrollment and study vaccination are acceptable provided there was no deterioration in the subject's chronic medical condition that necessitated a medication change, and there is no additional risk to the subject or interference with the evaluation of responses to study vaccination. Note: Topical, nasal, and inhaled medications (apart from steroids as outlined in the Subject Exclusion Criteria), herbals, vitamins, and supplements are permitted.
6. Oral temperature is less than 100.0 degrees Fahrenheit (37.8 degrees Celsius).
7. Pulse is 47 to 105 beats per minute (bpm), inclusive.
8. Systolic blood pressure (BP) is 85 to 150 mm Hg, inclusive.
9. Diastolic blood pressure (BP) is 55 to 95 mm Hg, inclusive.
10. Have acceptable screening laboratories within 28 days prior to enrollment

    * Screening labs include white blood cell (WBC), Hgb, platelet count, ANC, sodium, potassium, creatinine, albumin, total protein, PT, PTT, alanine aminotransferase (ALT). Blood Urea Nitrogen (BUN) will be obtained only if creatinine is above normal range.

      * Screening laboratory values that are outside the range of eligibility but are thought to be due to an acute condition or due to laboratory error may be repeated once.
11. Have normal screening laboratories for urine protein. Trace protein is acceptable.
12. Drug screen for opiates is negative.
13. Hemoglobin A1C (HgbA1C) < 6.3% at screening.
14. HIV 1/2 antibody negative.
15. HCV antibody negative.
16. HBsAg negative.
17. Women of childbearing potential, must be using an effective method of contraception from 30 days prior to the first study vaccination until 90 days after the second study vaccination.

    - Women of childbearing potential are not sterilized via tubal ligation, bilateral oophorectomy, hysterectomy, successful Essure(R) placement (permanent, non-surgical, non-hormonal sterilization) with history of documented radiological confirmation test at least 90 days after the procedure (or with use of another birth control method if history of confirmation test not confirmed), still menstruating, or < 1 year of the last menses if menopausal.

    -- Effective methods of contraception includes, but is not limited to, non-male sexual relationships, abstinence from sexual intercourse with a male partner, monogamous relationship with a vasectomized partner, male condoms with the use of applied spermicide, intrauterine devices, NuvaRing(R), and licensed hormonal methods such as implants, injectables or oral contraceptives ("the pill").
18. Women of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test within 24 hours prior to each study vaccination.
19. Women agree to not donate eggs (ova, oocytes) from the start of screening onwards until at least 90 days after the second vaccination.
20. Agrees not to participate in another clinical trial during the study period.
21. Agrees not to donate blood to a blood bank for 3 months after receiving the second study vaccine.

Exclusion Criteria:

1. Women who are pregnant, planning to become pregnant or lactating. - Includes breastfeeding or planning to breastfeed at any given time from the receipt of study vaccination through the 6-month trial period.
2. Known allergy or history of anaphylaxis, severe local or other serious adverse reactions to vaccines or vaccine products, or history of severe allergic reactions.

   - Includes a known allergy to egg, egg products and aminoglycosides or any of the constituents of the study vaccines [e.g., polysorbate 80, ethylenediaminetetraacetic acid (EDTA), L-histidine, tris (hydroxymethyl)-amino methane (THAM)).
3. Received an experimental agent within 3 months prior to Day 1, or expects to receive an experimental agent (other than from participation in this study) during the 6-month trial-reporting period.

   - Including vaccine, drug, biologic, device, blood product, or medication.
4. Received immunoglobulin or other blood product within 3 months before enrollment in this study.
5. Received any licensed live vaccine within 30 days prior to the first study vaccination through 30 days after the second study vaccination.
6. Received a licensed inactivated vaccine within 14 days prior to the first study vaccination through 14 days after the second study vaccination.
7. Has been vaccinated with an Ebola vaccine.
8. Has been diagnosed with Ebola disease, or exposed to Ebola virus including travel to West Africa in 2014-2016.

   - West Africa includes but is not limited to the countries of Guinea, Liberia, Mali, Nigeria, and Sierra Leone.
9. Known or suspected receipt of ChAd3-EBO-Z or other ChAd3-vectored vaccine.
10. Known or suspected receipt of an adenovirus serotype 5 (Ad5)-based vaccine.
11. Known or suspected receipt of any licensed or investigational small pox (vaccinia)-based vaccine.

    - Includes any MVA-based candidate vaccine (Imvamune or Imvanex), Dryvax, or Acam2000.
12. Has a typical vaccinia scar.
13. Confirmed Asplenia/Functional Asplenia.
14. A history of bleeding or clotting disorders.
15. Thyroidectomy or thyroid disease requiring medication during the last 12 months.
16. History of chronic urticaria (recurrent hives).
17. Individuals in whom the ability to observe possible local reactions at the eligible injection sites (left and right deltoid region) is, unacceptably obscured due to a physical condition or permanent body art.
18. Have an acute illness, as determined by the site PI or appropriate sub-investigator, within 72 hours prior to study vaccination.

    - An acute illness which is nearly resolved with only minor residual symptoms remaining is allowable if, in the opinion of the site PI or appropriate sub-investigator, the residual symptoms will not interfere with the ability to assess safety parameters as required by the protocol. Subjects may re-screen after an acute illness is resolved.
19. Any confirmed or suspected immunosuppressive or immunodeficient condition (including HIV infection) or use of anticancer chemotherapy or radiation therapy (cytotoxic) within 3 years prior to study vaccination
20. Administration of chronic (defined as more than 14 days) immunosuppressants or other immune modifying drugs within 6 months of receipt of study vaccine.
21. Have taken oral or parenteral (including intraarticular) corticosteroids of any dose within 30 days prior to study vaccination.
22. Have taken high-dose dose inhaled corticosteroids within 30 days prior to study vaccination.

    - High-dose defined using the inhaled high-dose reference chart.
23. Have a history of convulsions or encephalomyelitis within 90 days prior to study vaccination.
24. Current or past history of alcohol or drug abuse in the last 5 years.
25. Subjects with autoimmune disorders, chronic inflammatory disorders or neurological disorders with a potential autoimmune correlation.
26. Have any diagnosis, current or past, of schizophrenia, bipolar disease, or other psychiatric diagnosis that may interfere with subject compliance or safety evaluations.
27. Have been hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others within 10 years prior to study vaccination.
28. Have received any antiviral within 3 days of study vaccination
29. History of myocarditis, pericarditis, cardiomyopathy, transient ischemic attack or stroke, myocardial infarction, angina, coronary artery disease, congestive heart failure, clinically significant arrhythmia.

    - Including any arrhythmia requiring medication, treatment, or clinical follow-up.
30. Electrocardiogram (ECG) with clinically significant findings.

    - Clinically significant findings include the following:
    * Conduction disturbance (complete left or complete right bundle branch block or nonspecific intraventricular conduction disturbance with QRS = / > 120 ms, PR interval = / > 210 ms, any second- or third-degree atrioventricular block, or prolongation of the QT interval corrected according to Bazett's formula [QTcB] [> 450 ms]).
    * Significant repolarization (ST-segment or T-wave) abnormality.
    * Significant atrial or ventricular arrhythmia; frequent atrial or ventricular ectopy (e.g., frequent premature atrial contractions, 2 premature ventricular contractions in a row).
    * ST-elevation consistent with ischemia or evidence of past or evolving myocardial infarction
31. A diagnosis of Type I or II diabetes. (A history of isolated gestational diabetes is not an exclusion criterion).
32. Current employee or staff paid entirely or partially by the contract for this trial, or staff who are supervised by the PI or Sub-Investigators.
33. Any condition that would, in the opinion of the Site Investigator or appropriate sub-investigator, is a contraindication to study participation.

    * Including acute or chronic (persisting for at least 90 days) clinically significant medical disease or condition, that would place the subject at an unacceptable risk of injury, render the subject unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the subject's successful completion of the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2020-01-14 (Actual); Study Completion 2020-01-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center Vaccine Research Center, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were males and non-pregnant females in good health, aged 19 to 45, and recruited from the community at large at the participating site. Participants were enrolled between 12NOV2018 to 10JUL2019.
Groups:
- ChAd3-EBO-Z + Placebo: ChAd3-EBO-Z (2 x 10^11 virus particles (vp)) intramuscularly into the deltoid on Day 1 and placebo intramuscularly into the opposite arm on Day 8 (+2). All participants in all Study Arms received the same product (ChAd3-EBO-Z) at Day 1.
  ChAd3-EBO-Z: Zaire ebolavirus vaccine administered by an IM injection into the deltoid as a single dose of 2 x 10^11 virus particles (vp)).
  Placebo: 0.5 mL normal saline administered via IM injection into the deltoid.
- ChAd3-EBO-Z + ChAd3-EBO-Z: ChAd3-EBO-Z (2 x 10^11 virus particles (vp)) intramuscularly into the deltoid on Day 1 and ChAd3-EBO-Z (2 x 10^11 vp) intramuscularly into the opposite arm on Day 8 (+2). All participants in all Study Arms received the same product (ChAd3-EBO-Z) at Day 1.
  ChAd3-EBO-Z: Zaire ebolavirus vaccine administered by an IM injection into the deltoid as a single dose of 2 x 10^11 virus particles (vp)).
- ChAd3-EBO-Z + MVA- BN-Filo: ChAd3-EBO-Z (2 x 10^11 virus particles (vp)) intramuscularly into the deltoid on Day 1 and MVA-BN-Filo (1 x 10^8 Infectious Units (IU)) intramuscularly into the opposite arm on Day 8 (+2). All participants in all Study Arms received the same product (ChAd3-EBO-Z) at Day 1.
  ChAd3-EBO-Z: Zaire ebolavirus vaccine administered by an IM injection into the deltoid as a single dose of 2 x 10^11 virus particles (vp)).
  MVA Multi-Filo Ebola Vaccine: A booster vaccination of replication defective MVA-BN-Filo administered by an IM injection into the deltoid as a single dose of 1 x 10^8 Infectious Units (IU).
Period: Overall Study
Arm/Group | ChAd3-EBO-Z + Placebo | ChAd3-EBO-Z + ChAd3-EBO-Z | ChAd3-EBO-Z + MVA- BN-Filo
Started | 22 | 20 | 19
Completed | 21 | 19 | 19
Not Completed | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Ineligible at baseline | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- ChAd3-EBO-Z + Placebo: ChAd3-EBO-Z (2 x 10^11 virus particles (vp)) intramuscularly into the deltoid on Day 1 and placebo intramuscularly into the opposite arm on Day 8.
  ChAd3-EBO-Z: Zaire ebolavirus vaccine administered by an IM injection into the deltoid as a single dose of 2 x 10^11 virus particles (vp)).
  Placebo: 0.5 mL normal saline administered via IM injection into the deltoid.
- ChAd3-EBO-Z + ChAd3-EBO-Z: ChAd3-EBO-Z (2 x 10^11 virus particles (vp)) intramuscularly into the deltoid on Day 1 and ChAd3-EBO-Z (2 x 10^11 vp) intramuscularly into the opposite arm on Day 8.
  ChAd3-EBO-Z: Zaire ebolavirus vaccine administered by an IM injection into the deltoid as a single dose of 2 x 10^11 virus particles (vp)).
- ChAd3-EBO-Z + MVA- BN-Filo: ChAd3-EBO-Z (2 x 10^11 virus particles (vp)) intramuscularly into the deltoid on Day 1 and MVA-BN-Filo (1 x 10^8 Infectious Units (IU)) intramuscularly into the opposite arm on Day 8.
  ChAd3-EBO-Z: Zaire ebolavirus vaccine administered by an IM injection into the deltoid as a single dose of 2 x 10^11 virus particles (vp)).
  MVA Multi-Filo Ebola Vaccine: A booster vaccination of replication defective MVA-BN-Filo administered by an IM injection into the deltoid as a single dose of 1 x 10^8 Infectious Units (IU).
- Total: Total of all reporting groups
Arm/Group | ChAd3-EBO-Z + Placebo | ChAd3-EBO-Z + ChAd3-EBO-Z | ChAd3-EBO-Z + MVA- BN-Filo | Total
Number analyzed (Participants) | 22 | 20 | 19 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 22 | 20 | 19 | 61
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.8 (7.8) | 26.8 (5.3) | 31.4 (7.6) | 30.8 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 13 | 35
  Male | 11 | 9 | 6 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 2 | 6
  Not Hispanic or Latino | 19 | 19 | 17 | 55
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 0 | 2 | 5
  White | 16 | 19 | 15 | 50
  More than one race | 2 | 1 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 22 | 20 | 19 | 61
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.35 (3.96) | 25.19 (3.77) | 25.49 (4.06) | 25.70 (3.90)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Safety Laboratory Adverse Events
Description: Laboratory parameters include white blood cells (WBC), hemoglobin, platelet count, absolute neutrophil count, alanine aminotransferase (ALT), creatinine, sodium, potassium and blood urea nitrogen (BUN). Thresholds for adverse events were considered as WBC <= 4.4 K/mcL or >=13.1 K/mcL (18 to <21 years) or <= 4.4 K/mcL or >= 11.1 K/mcL (>=21 years), hemoglobin <= 11.6 g/dL (female) or <= 13.2 g/dL (male), platelet count <= 134 K/mcL or >= 467 K/mcL, absolute neutrophil count <1.8 K/mcL or <=0.7 K/mcL (benign ethnic neutropenia), ALT >= 50 unit/L, creatinine >= 0.81 mg/dL (female) or >= 1.11 mg/dL (male), sodium <= 135 mmol/L or >= 146 mmol/L, potassium <= 3.4 mmol/L or >= 5.2 mmol/L and BUN >= 24 mg/dL. If baseline clinical labs fell within Mild range, then a laboratory AE was reported only if the value changed such that it fell into Moderate range or higher when subsequent safety laboratory testing was done.
Time Frame: Day 1 to approximately 28 Days Post Second Vaccination
Population: Safety Population: includes all participants who received at least one study vaccination.
Measure: Count of Participants; unit: Participants
Groups:
- ChAd3-EBO-Z + Placebo: ChAd3-EBO-Z (2 x 10^11 virus particles (vp)) intramuscularly into the deltoid on Day 1 and placebo intramuscularly into the opposite arm on Day 8.
- ChAd3-EBO-Z + ChAd3-EBO-Z: ChAd3-EBO-Z (2 x 10^11 virus particles (vp)) intramuscularly into the deltoid on Day 1 and ChAd3-EBO-Z (2 x 10^11 vp) intramuscularly into the opposite arm on Day 8.
- ChAd3-EBO-Z + MVA- BN-Filo: ChAd3-EBO-Z (2 x 10^11 virus particles (vp)) intramuscularly into the deltoid on Day 1 and MVA-BN-Filo (1 x 10^8 Infectious Units (IU)) intramuscularly into the opposite arm on Day 8.
Arm/Group | ChAd3-EBO-Z + Placebo | ChAd3-EBO-Z + ChAd3-EBO-Z | ChAd3-EBO-Z + MVA- BN-Filo
Number analyzed (Participants) | 21 | 20 | 19
Participants
  WBC | 2 | 5 | 4
  Hemoglobin | 2 | 6 | 2
  Platelet count | 1 | 1 | 1
  Absolute neutrophil count | 1 | 5 | 3
  ALT | 1 | 2 | 1
  Creatinine | 2 | 1 | 2
  Sodium | 1 | 0 | 0
  Potassium | 1 | 0 | 0
  BUN | 0 | 0 | 0

2. Primary Outcome: Number of Participants Reporting Serious Adverse Events (SAEs)
Description: SAEs included any AE that resulted in death, a life-threatening event, an inpatient hospitalization or prolongation of existing hospitalization, a persistent/significant disability/incapacity, or a congenital anomaly/birth defect.
Time Frame: Day 1 to Day 182
Population: Safety Population: includes all participants who received at least one study vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | ChAd3-EBO-Z + Placebo | ChAd3-EBO-Z + ChAd3-EBO-Z | ChAd3-EBO-Z + MVA- BN-Filo
Number analyzed (Participants) | 21 | 20 | 19
Participants | 0 | 0 | 0

3. Primary Outcome: Number of Participants Reporting Solicited Local Reactogenicity
Description: Local reactogenicity solicited on a memory aid provided to participants included pain, tenderness, erythema (redness) (functional grade based on interference with daily activities), induration (hardness/swelling) (functional grade), ecchymosis (bruising) (functional grade), pruritus (itching), erythema (redness) (any measured value), induration (hardness/swelling) (any measured value), ecchymosis (bruising) (any measured value). Participants are considered reporting the local reactogenicity if they reported mild or greater severity at any time during the 7 days post-vaccination.
Time Frame: Day 1 to Day 8 Post First Vaccination
Population: Safety Population: includes all participants who received at least one study vaccination. All participants in all Study Arms received the same product (ChAd3-EBO-Z) at Day 1.
Measure: Count of Participants; unit: Participants
Groups:
- ChAd3-EBO-Z + MVABN-Filo: ChAd3-EBO-Z (2 x 10^11 virus particles (vp)) intramuscularly into the deltoid on Day 1 and MVA-BN-Filo (1 x 10^8 Infectious Units (IU)) intramuscularly into the opposite arm on Day 8.
Arm/Group | ChAd3-EBO-Z + Placebo | ChAd3-EBO-Z + ChAd3-EBO-Z | ChAd3-EBO-Z + MVABN-Filo
Number analyzed (Participants) | 21 | 20 | 19
Participants
  Any Local Symptom | 20 | 20 | 18
  Pain | 13 | 17 | 14
  Tenderness | 17 | 19 | 15
  Pruritus | 1 | 0 | 0
  Ecchymosis (Functional Grade) | 0 | 2 | 2
  Ecchymosis (Measurement Grade) | 0 | 2 | 2
  Erythema (Functional Grade) | 7 | 11 | 11
  Erythema (Measurement Grade) | 7 | 11 | 11
  Induration (Functional Grade) | 6 | 7 | 5
  Induration (Measurement Grade) | 6 | 7 | 5

4. Primary Outcome: Number of Participants Reporting Solicited Local Reactogenicity
Description: as for outcome 3
Time Frame: Day 1 to Day 8 Post Second Vaccination
Population: Safety Population Subset: includes all participants who received the first and second study vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | ChAd3-EBO-Z + Placebo | ChAd3-EBO-Z + ChAd3-EBO-Z | ChAd3-EBO-Z + MVA- BN-Filo
Number analyzed (Participants) | 17 | 17 | 18
Participants
  Any Local Symptom | 6 | 17 | 13
  Pain | 1 | 13 | 5
  Tenderness | 3 | 15 | 12
  Pruritus | 0 | 1 | 1
  Ecchymosis (Functional Grade) | 0 | 0 | 0
  Ecchymosis (Measurement Grade) | 0 | 0 | 0
  Erythema (Functional Grade) | 5 | 7 | 6
  Erythema (Measurement Grade) | 5 | 7 | 6
  Induration (Functional Grade) | 0 | 3 | 1
  Induration (Measurement Grade) | 0 | 3 | 1

5. Primary Outcome: Number of Participants Reporting Solicited Local Reactogenicity
Description: Local reactogenicity solicited on a memory aid provided to participants included pain, tenderness, erythema (redness) (functional grade based on interference with daily activities), induration (hardness/swelling) (functional grade), ecchymosis (bruising) (functional grade), pruritus (itching), erythema (redness) (any measured value), induration (hardness/swelling) (any measured value), ecchymosis (bruising) (any measured value). Subjects are considered reporting the local reactogenicity if they reported mild or greater severity at any time during the 7 days post-vaccination.
Time Frame: Day 1 to Day 15
Population: Safety Population: includes all participants who received at least one study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | ChAd3-EBO-Z + Placebo | ChAd3-EBO-Z + ChAd3-EBO-Z | ChAd3-EBO-Z + MVA- BN-Filo
Number analyzed (Participants) | 21 | 20 | 19
Participants
  Any Local Symptom | 20 | 20 | 18
  Pain | 13 | 18 | 14
  Tenderness | 17 | 19 | 15
  Pruritus | 1 | 1 | 1
  Ecchymosis (functional grade) | 0 | 2 | 2
  Ecchymosis (measurement grade) | 0 | 2 | 2
  Erythema (functional grade) | 10 | 11 | 12
  Erythema (measurement grade) | 10 | 11 | 12
  Induration (functional grade) | 6 | 8 | 5
  Induration (measurement grade) | 6 | 8 | 5

6. Primary Outcome: Number of Participants Reporting Solicited Systemic Reactogenicity
Description: Systemic reactogenicity solicited on a memory aid provided to participants included feverishness (chills/shivering/sweating), malaise (general unwell feeling), fatigue (tiredness), myalgia (body aches/muscular pain not at injection site), headache, nausea, loss of appetite, and elevated oral temperature. Participants are considered reporting the systemic reactogenicity if they reported mild or greater severity at any time during the 7 days post-vaccination.
Time Frame: Day 1 to Day 8 Post First Vaccination
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | ChAd3-EBO-Z + Placebo | ChAd3-EBO-Z + ChAd3-EBO-Z | ChAd3-EBO-Z + MVABN-Filo
Number analyzed (Participants) | 21 | 20 | 19
Participants
  Any Systemic Symptom | 20 | 20 | 15
  Elevated Oral Temperature | 11 | 9 | 9
  Feverishness | 15 | 14 | 13
  Malaise | 13 | 17 | 13
  Fatigue | 17 | 15 | 13
  Myalgia | 17 | 17 | 12
  Headache | 10 | 10 | 12
  Nausea | 6 | 9 | 3
  Loss of Appetite | 4 | 9 | 8

7. Primary Outcome: Number of Participants Reporting Solicited Systemic Reactogenicity
Description: as for outcome 6
Time Frame: Day 1 to Day 8 Post Second Vaccination
Population: Safety Population Subset: includes all participants who received the first and second study vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | ChAd3-EBO-Z + Placebo | ChAd3-EBO-Z + ChAd3-EBO-Z | ChAd3-EBO-Z + MVA- BN-Filo
Number analyzed (Participants) | 17 | 17 | 18
Participants
  Any Systemic Symptom | 8 | 14 | 6
  Elevated Oral Temperature | 0 | 8 | 0
  Feverishness | 3 | 11 | 1
  Malaise | 3 | 14 | 1
  Fatigue | 7 | 14 | 3
  Myalgia | 3 | 11 | 4
  Headache | 7 | 9 | 4
  Nausea | 2 | 4 | 1
  Loss of Appetite | 3 | 7 | 0

8. Primary Outcome: Number of Participants Reporting Solicited Systemic Reactogenicity
Description: as for outcome 6
Time Frame: Day 1 to Day 15
Population: Safety Population: includes all participants who received at least one study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | ChAd3-EBO-Z + Placebo | ChAd3-EBO-Z + ChAd3-EBO-Z | ChAd3-EBO-Z + MVA- BN-Filo
Number analyzed (Participants) | 21 | 20 | 19
Participants
  Any Systemic Symptom | 20 | 20 | 15
  Elevated Oral Temperature | 11 | 12 | 9
  Feverishness | 18 | 16 | 13
  Malaise | 14 | 19 | 13
  Fatigue | 18 | 19 | 13
  Myalgia | 17 | 20 | 12
  Headache | 13 | 13 | 12
  Nausea | 7 | 10 | 3
  Loss of Appetite | 6 | 12 | 8

9. Primary Outcome: Number of Participants Reporting Vaccine-related Medically Attended Adverse Events (MAAEs)
Description: Vaccine-related MAAEs include any AEs for which the participant received medical attention, defined as hospitalization, an emergency room visit, or an otherwise unscheduled visit to or from medical personnel for any reason for which there is evidence to suggest a causal relationship between the study product and the adverse event.
Time Frame: Day 1 to Day 182
Population: Safety Population: includes all participants who received at least one study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | ChAd3-EBO-Z + Placebo | ChAd3-EBO-Z + ChAd3-EBO-Z | ChAd3-EBO-Z + MVA- BN-Filo
Number analyzed (Participants) | 21 | 20 | 19
Participants | 0 | 0 | 0

10. Primary Outcome: Number of Participants Reporting Vaccine-related Unsolicited Adverse Events (AEs)
Description: Vaccine-related unsolicited AEs include any untoward medical occurrence in a participant for which there is evidence to suggest a causal relationship between the study product and the adverse event.
Time Frame: Day 1 to approximately 28 Days Post Second Vaccination
Population: Safety Population: includes all participants who received at least one study vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | ChAd3-EBO-Z + Placebo | ChAd3-EBO-Z + ChAd3-EBO-Z | ChAd3-EBO-Z + MVA- BN-Filo
Number analyzed (Participants) | 21 | 20 | 19
Participants
  Any SOC | 4 | 10 | 4
  Lymphadenopathy | 1 | 1 | 1
  Tachycardia | 0 | 1 | 0
  Diarrhea | 0 | 1 | 0
  Vomiting | 1 | 2 | 1
  Chest discomfort | 0 | 1 | 0
  Blood pressure diastolic decreased | 0 | 0 | 1
  Transaminases increased | 0 | 1 | 0
  Dehydration | 0 | 1 | 0
  Back pain | 0 | 1 | 0
  Muscle spasms | 0 | 0 | 1
  Dizziness | 0 | 1 | 0
  Sinus headache | 1 | 0 | 0
  Taste disorder | 0 | 1 | 0
  Cough | 1 | 0 | 0
  Oropharyngeal pain | 1 | 0 | 0
  Sinus congestion | 0 | 1 | 0
  Acne | 0 | 1 | 0
  Ecchymosis | 0 | 1 | 0
  Rash | 0 | 1 | 0

11. Primary Outcome: Number of Participants by Severity of Clinical Safety Laboratory Adverse Events - White Blood Cells
Description: Thresholds for adverse events were considered as WBC 2.5 - 4.4 K/mcL or 13.1 - 15.0 K/mcL (18 to <21 years) or 2.5 - 4.4 K/mcL or 11.1 - 15.0 (>=21 years) (mild), 1.5 - 2.4 K/mcL or 15.1 - 20.0 K/mcL (moderate), <1.5 K/mcL or >20.0 K/mcL (severe). If baseline clinical labs fell within mild range, then a laboratory AE was reported only if the value changed such that it fell into moderate range or higher when subsequent safety laboratory testing was done.
Time Frame: Day 1 to approximately 28 Days Post Second Vaccination
Population: Safety Population: includes all Participants who received at least one study vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | ChAd3-EBO-Z + Placebo | ChAd3-EBO-Z + ChAd3-EBO-Z | ChAd3-EBO-Z + MVA- BN-Filo
Number analyzed (Participants) | 21 | 20 | 19
Participants
  Day 8 (Second Vaccination): None | 19 | 18 | 17
  Day 8 (Second Vaccination): Mild (low) | 2 | 2 | 2
  Day 8 (Second Vaccination): Mild (high) | 0 | 0 | 0
  Day 8 (Second Vaccination): Moderate (low) | 0 | 0 | 0
  Day 8 (Second Vaccination): Moderate (high) | 0 | 0 | 0
  Day 8 (Second Vaccination): Severe | 0 | 0 | 0
  Day 8 (Second Vaccination): Missing | 0 | 0 | 0
  Day 8 Post-Second Vaccination: None | 20 | 17 | 18
  Day 8 Post-Second Vaccination: Mild (low) | 1 | 1 | 0
  Day 8 Post-Second Vaccination: Mild (high) | 0 | 1 | 0
  Day 8 Post-Second Vaccination: Moderate (low) | 0 | 0 | 0
  Day 8 Post-Second Vaccination: Moderate (high) | 0 | 0 | 0
  Day 8 Post-Second Vaccination: Severe | 0 | 0 | 0
  Day 8 Post-Second Vaccination: Missing | 0 | 1 | 1
  Day 22 Post-Second Vaccination: None | 20 | 16 | 17
  Day 22 Post-Second Vaccination: Mild (low) | 1 | 2 | 2
  Day 22 Post-Second Vaccination: Mild (high) | 0 | 1 | 0
  Day 22 Post-Second Vaccination: Moderate (low) | 0 | 0 | 0
  Day 22 Post-Second Vaccination: Moderate (high) | 0 | 0 | 0
  Day 22 Post-Second Vaccination: Severe | 0 | 0 | 0
  Day 22 Post-Second Vaccination: Missing | 0 | 1 | 0
  Day 29 Post-Second Vaccination: None | 19 | 17 | 19
  Day 29 Post-Second Vaccination: Mild (low) | 2 | 2 | 0
  Day 29 Post-Second Vaccination: Mild (high) | 0 | 0 | 0
  Day 29 Post-Second Vaccination: Moderate (low) | 0 | 0 | 0
  Day 29 Post-Second Vaccination: Moderate (high) | 0 | 0 | 0
  Day 29 Post-Second Vaccination: Severe | 0 | 0 | 0
  Day 29 Post-Second Vaccination: Missing | 0 | 1 | 0
  Max Severity Post Baseline: None | 19 | 15 | 15
  Max Severity Post Baseline: Mild (low) | 2 | 4 | 4
  Max Severity Post Baseline: Mild (high) | 0 | 1 | 0
  Max Severity Post Baseline: Moderate (low) | 0 | 0 | 0
  Max Severity Post Baseline: Moderate (high) | 0 | 0 | 0
  Max Severity Post Baseline: Severe | 0 | 0 | 0
  Max Severity Post Baseline: Missing | 0 | 0 | 0

12. Primary Outcome: Number of Participants by Severity of Clinical Safety Laboratory Adverse Events - Hemoglobin
Description: Thresholds for adverse events were considered as hemoglobin 10.1 - 11.6 g/dL (female) or 11.0 - 13.2 (male) (mild), 8.5 - 10 g/dL (female) or 9.5 - 10.9 g/dL (male) (moderate), <8.5 g/dL (female) or <9.5 g/dL (male) (severe). If baseline clinical labs fell within mild range, then a laboratory AE was reported only if the value changed such that it fell into moderate range or higher when subsequent safety laboratory testing was done.
Time Frame: Day 1 to approximately 28 Days Post Second Vaccination
Population: Safety Population: includes all participants who received at least one study vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | ChAd3-EBO-Z + Placebo | ChAd3-EBO-Z + ChAd3-EBO-Z | ChAd3-EBO-Z + MVA- BN-Filo
Number analyzed (Participants) | 21 | 20 | 19
Participants
  Day 8 (Second Vaccination): None | 19 | 20 | 18
  Day 8 (Second Vaccination): Mild | 2 | 0 | 1
  Day 8 (Second Vaccination): Moderate | 0 | 0 | 0
  Day 8 (Second Vaccination): Severe | 0 | 0 | 0
  Day 8 (Second Vaccination): Missing | 0 | 0 | 0
  Day 8 Post-Second Vaccination: None | 19 | 14 | 17
  Day 8 Post-Second Vaccination: Mild | 2 | 5 | 1
  Day 8 Post-Second Vaccination: Moderate | 0 | 0 | 0
  Day 8 Post-Second Vaccination: Severe | 0 | 0 | 0
  Day 8 Post-Second Vaccination: Missing | 0 | 1 | 1
  Day 22 Post-Second Vaccination: None | 19 | 15 | 17
  Day 22 Post-Second Vaccination: Mild | 2 | 4 | 2
  Day 22 Post-Second Vaccination: Moderate | 0 | 0 | 0
  Day 22 Post-Second Vaccination: Severe | 0 | 0 | 0
  Day 22 Post-Second Vaccination: Missing | 0 | 1 | 0
  Day 29 Post-Second Vaccination: None | 19 | 16 | 18
  Day 29 Post-Second Vaccination: Mild | 1 | 3 | 1
  Day 29 Post-Second Vaccination: Moderate | 1 | 0 | 0
  Day 29 Post-Second Vaccination: Severe | 0 | 0 | 0
  Day 29 Post-Second Vaccination: Missing | 0 | 1 | 0
  Max Severity Post Baseline: None | 19 | 14 | 17
  Max Severity Post Baseline: Mild | 1 | 6 | 2
  Max Severity Post Baseline: Moderate | 1 | 0 | 0
  Max Severity Post Baseline: Severe | 0 | 0 | 0
  Max Severity Post Baseline: Missing | 0 | 0 | 0

13. Primary Outcome: Number of Participants by Severity of Clinical Safety Laboratory Adverse Events - Platelet Count
Description: Thresholds for adverse events were considered as platelet count 125 - 134 K/mcL or 467 - 517 K/mcL (mild), 100 - 124 K/mcL or 518 - 750 K/mcL (moderate), <100 K/mcL or >750 K/mcL (severe). If baseline clinical labs fell within mild range, then a laboratory AE was reported only if the value changed such that it fell into moderate range or higher when subsequent safety laboratory testing was done.
Time Frame: Day 1 to approximately 28 Days Post Second Vaccination
Population: Safety Population: includes all participants who received at least one study vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | ChAd3-EBO-Z + Placebo | ChAd3-EBO-Z + ChAd3-EBO-Z | ChAd3-EBO-Z + MVA- BN-Filo
Number analyzed (Participants) | 21 | 20 | 19
Participants
  Day 8 (Second Vaccination): None | 21 | 20 | 19
  Day 8 (Second Vaccination): Mild (low) | 0 | 0 | 0
  Day 8 (Second Vaccination): Mild (high) | 0 | 0 | 0
  Day 8 (Second Vaccination): Moderate (low) | 0 | 0 | 0
  Day 8 (Second Vaccination): Severe (low or high) | 0 | 0 | 0
  Day 8 (Second Vaccination): Missing | 0 | 0 | 0
  Day 8 Post-Second Vaccination: None | 21 | 19 | 18
  Day 8 Post-Second Vaccination: Mild (low) | 0 | 0 | 0
  Day 8 Post-Second Vaccination: Mild (high) | 0 | 0 | 0
  Day 8 Post-Second Vaccination: Moderate (low) | 0 | 0 | 0
  Day 8 Post-Second Vaccination: Severe (low or high) | 0 | 0 | 0
  Day 8 Post-Second Vaccination: Missing | 0 | 1 | 1
  Day 22 Post-Second Vaccination: None | 21 | 19 | 19
  Day 22 Post-Second Vaccination: Mild (low) | 0 | 0 | 0
  Day 22 Post-Second Vaccination: Mild (high) | 0 | 0 | 0
  Day 22 Post-Second Vaccination: Moderate (low) | 0 | 0 | 0
  Day 22 Post-Second Vaccination: Severe (low or high) | 0 | 0 | 0
  Day 22 Post-Second Vaccination: Missing | 0 | 1 | 0
  Day 29 Post-Second Vaccination: None | 21 | 18 | 19
  Day 29 Post-Second Vaccination: Mild (low) | 0 | 1 | 0
  Day 29 Post-Second Vaccination: Mild (high) | 0 | 0 | 0
  Day 29 Post-Second Vaccination: Moderate (low) | 0 | 0 | 0
  Day 29 Post-Second Vaccination: Severe (low or high) | 0 | 0 | 0
  Day 29 Post-Second Vaccination: Missing | 0 | 1 | 0
  Max Severity Post Baseline: None | 20 | 19 | 18
  Max Severity Post Baseline: Mild (low) | 0 | 1 | 0
  Max Severity Post Baseline: Mild (high) | 1 | 0 | 0
  Max Severity Post Baseline: Moderate (low) | 0 | 0 | 1
  Max Severity Post Baseline: Severe (low or high) | 0 | 0 | 0
  Max Severity Post Baseline: Missing | 0 | 0 | 0

14. Primary Outcome: Number of Participants by Severity of Clinical Safety Laboratory Adverse Events - Absolute Neutrophil Count
Description: Thresholds for adverse events were considered as absolute neutrophil count 1.5 - <1.8 K/mcL or 0.6 - 0.7 K/mcL (benign ethnic neutropenia) (mild), 1.0 - <1.5 K/mcL or 0.4 - 0.5 K/mcL (benign ethnic neutropenia) (moderate), <1.0 K/mcL or <0.4 K/mcL (benign ethnic neutropenia) (severe). If baseline clinical labs fell within mild range, then a laboratory AE was reported only if the value changed such that it fell into moderate range or higher when subsequent safety laboratory testing was done.
Time Frame: Day 1 to approximately 28 Days Post Second Vaccination
Population: Safety Population: includes all participants who received at least one study vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | ChAd3-EBO-Z + Placebo | ChAd3-EBO-Z + ChAd3-EBO-Z | ChAd3-EBO-Z + MVA- BN-Filo
Number analyzed (Participants) | 21 | 20 | 19
Participants
  Day 8 (Second Vaccination): None | 19 | 17 | 17
  Day 8 (Second Vaccination): Mild | 0 | 2 | 0
  Day 8 (Second Vaccination): Moderate | 1 | 1 | 2
  Day 8 (Second Vaccination): Severe | 0 | 0 | 0
  Day 8 (Second Vaccination): Missing | 1 | 0 | 0
  Day 8 Post-Second Vaccination: None | 21 | 19 | 17
  Day 8 Post-Second Vaccination: Mild | 0 | 0 | 1
  Day 8 Post-Second Vaccination: Moderate | 0 | 0 | 0
  Day 8 Post-Second Vaccination: Severe | 0 | 0 | 0
  Day 8 Post-Second Vaccination: Missing | 0 | 1 | 1
  Day 22 Post-Second Vaccination: None | 21 | 17 | 18
  Day 22 Post-Second Vaccination: Mild | 0 | 1 | 1
  Day 22 Post-Second Vaccination: Moderate | 0 | 1 | 0
  Day 22 Post-Second Vaccination: Severe | 0 | 0 | 0
  Day 22 Post-Second Vaccination: Missing | 0 | 1 | 0
  Day 29 Post-Second Vaccination: None | 21 | 17 | 18
  Day 29 Post-Second Vaccination: Mild | 0 | 2 | 1
  Day 29 Post-Second Vaccination: Moderate | 0 | 0 | 0
  Day 29 Post-Second Vaccination: Severe | 0 | 0 | 0
  Day 29 Post-Second Vaccination: Missing | 0 | 1 | 0
  Max Severity Post Baseline: None | 20 | 15 | 16
  Max Severity Post Baseline: Mild | 0 | 3 | 1
  Max Severity Post Baseline: Moderate | 1 | 2 | 2
  Max Severity Post Baseline: Severe | 0 | 0 | 0
  Max Severity Post Baseline: Missing | 0 | 0 | 0

15. Primary Outcome: Number of Participants by Severity of Clinical Safety Laboratory Adverse Events - ALT
Description: Thresholds for adverse events were considered as 50 - 123 unit/L (mild), 124 - 245 unit/L (moderate), >245 unit/L (severe). If baseline clinical labs fell within mild range, then a laboratory AE was reported only if the value changed such that it fell into moderate range or higher when subsequent safety laboratory testing was done.
Time Frame: Day 1 to approximately 28 Days Post Second Vaccination
Population: Safety Population: includes all participants who received at least one study vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | ChAd3-EBO-Z + Placebo | ChAd3-EBO-Z + ChAd3-EBO-Z | ChAd3-EBO-Z + MVA- BN-Filo
Number analyzed (Participants) | 21 | 20 | 19
Participants
  Day 8 (Second Vaccination): None | 20 | 20 | 19
  Day 8 (Second Vaccination): Mild | 1 | 0 | 0
  Day 8 (Second Vaccination): Moderate | 0 | 0 | 0
  Day 8 (Second Vaccination): Severe | 0 | 0 | 0
  Day 8 (Second Vaccination): Missing | 0 | 0 | 0
  Day 8 Post-Second Vaccination: None | 20 | 19 | 17
  Day 8 Post-Second Vaccination: Mild | 1 | 0 | 1
  Day 8 Post-Second Vaccination: Moderate | 0 | 0 | 0
  Day 8 Post-Second Vaccination: Severe | 0 | 0 | 0
  Day 8 Post-Second Vaccination: Missing | 0 | 1 | 1
  Day 22 Post-Second Vaccination: None | 21 | 17 | 19
  Day 22 Post-Second Vaccination: Mild | 0 | 1 | 0
  Day 22 Post-Second Vaccination: Moderate | 0 | 1 | 0
  Day 22 Post-Second Vaccination: Severe | 0 | 0 | 0
  Day 22 Post-Second Vaccination: Missing | 0 | 1 | 0
  Day 29 Post-Second Vaccination: None | 21 | 18 | 18
  Day 29 Post-Second Vaccination: Mild | 0 | 1 | 1
  Day 29 Post-Second Vaccination: Moderate | 0 | 0 | 0
  Day 29 Post-Second Vaccination: Severe | 0 | 0 | 0
  Day 29 Post-Second Vaccination: Missing | 0 | 1 | 0
  Max Severity Post Baseline: None | 20 | 18 | 18
  Max Severity Post Baseline: Mild | 1 | 1 | 1
  Max Severity Post Baseline: Moderate | 0 | 1 | 0
  Max Severity Post Baseline: Severe | 0 | 0 | 0
  Max Severity Post Baseline: Missing | 0 | 0 | 0

16. Primary Outcome: Number of Participants by Severity of Clinical Safety Laboratory Adverse Events - Creatinine (Increase)
Description: Thresholds for adverse events were considered as creatinine 0.81 - 1.70 mg/dL (female) or 1.11 - 1.70 mg/dL (male) (mild), 1.71 - 2.00 mg/dL (moderate), >2.00 mg/dL (severe). If baseline clinical labs fell within mild range, then a laboratory AE was reported only if the value changed such that it fell into moderate range or higher when subsequent safety laboratory testing was done.
Time Frame: Day 1 to approximately 28 Days Post Second Vaccination
Population: Safety Population: includes all participants who received at least one study vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | ChAd3-EBO-Z + Placebo | ChAd3-EBO-Z + ChAd3-EBO-Z | ChAd3-EBO-Z + MVA- BN-Filo
Number analyzed (Participants) | 21 | 20 | 19
Participants
  Day 8 (Second Vaccination): None | 21 | 19 | 19
  Day 8 (Second Vaccination): Mild | 0 | 1 | 0
  Day 8 (Second Vaccination): Moderate | 0 | 0 | 0
  Day 8 (Second Vaccination): Severe | 0 | 0 | 0
  Day 8 (Second Vaccination): Missing | 0 | 0 | 0
  Day 8 Post-Second Vaccination: None | 20 | 19 | 16
  Day 8 Post-Second Vaccination: Mild | 1 | 0 | 2
  Day 8 Post-Second Vaccination: Moderate | 0 | 0 | 0
  Day 8 Post-Second Vaccination: Severe | 0 | 0 | 0
  Day 8 Post-Second Vaccination: Missing | 0 | 1 | 1
  Day 22 Post-Second Vaccination: None | 20 | 18 | 19
  Day 22 Post-Second Vaccination: Mild | 1 | 1 | 0
  Day 22 Post-Second Vaccination: Moderate | 0 | 0 | 0
  Day 22 Post-Second Vaccination: Severe | 0 | 0 | 0
  Day 22 Post-Second Vaccination: Missing | 0 | 1 | 0
  Day 29 Post-Second Vaccination: None | 19 | 19 | 19
  Day 29 Post-Second Vaccination: Mild | 2 | 0 | 0
  Day 29 Post-Second Vaccination: Moderate | 0 | 0 | 0
  Day 29 Post-Second Vaccination: Severe | 0 | 0 | 0
  Day 29 Post-Second Vaccination: Missing | 0 | 1 | 0
  Max Severity Post Baseline: None | 19 | 19 | 17
  Max Severity Post Baseline: Mild | 2 | 1 | 2
  Max Severity Post Baseline: Moderate | 0 | 0 | 0
  Max Severity Post Baseline: Severe | 0 | 0 | 0
  Max Severity Post Baseline: Missing | 0 | 0 | 0

17. Primary Outcome: Number of Participants by Severity of Clinical Safety Laboratory Adverse Events - Sodium
Description: Thresholds for adverse events were considered as sodium 130 - 135 mmol/L or 146 - 150 mmol/L (mild), 123 - 129 mmol/L or 151 - 157 mmol/L (moderate), <123 mmol/L or >157 mmol/L (severe). If baseline clinical labs fell within mild range, then a laboratory AE was reported only if the value changed such that it fell into moderate range or higher when subsequent safety laboratory testing was done.
Time Frame: Day 1 to approximately 28 Days Post Second Vaccination
Population: Safety Population: includes all participants who received at least one study vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | ChAd3-EBO-Z + Placebo | ChAd3-EBO-Z + ChAd3-EBO-Z | ChAd3-EBO-Z + MVA- BN-Filo
Number analyzed (Participants) | 21 | 20 | 19
Participants
  Day 8 (Second Vaccination): None | 21 | 20 | 19
  Day 8 (Second Vaccination): Mild (low) | 0 | 0 | 0
  Day 8 (Second Vaccination): Mild (high) | 0 | 0 | 0
  Day 8 (Second Vaccination): Moderate (low or high) | 0 | 0 | 0
  Day 8 (Second Vaccination): Severe (low or high) | 0 | 0 | 0
  Day 8 (Second Vaccination): Missing | 0 | 0 | 0
  Day 8 Post-Second Vaccination: None | 21 | 19 | 18
  Day 8 Post-Second Vaccination: Mild (low) | 0 | 0 | 0
  Day 8 Post-Second Vaccination: Mild (high) | 0 | 0 | 0
  Day 8 Post-Second Vaccination: Moderate (low or high) | 0 | 0 | 0
  Day 8 Post-Second Vaccination: Severe (low or high) | 0 | 0 | 0
  Day 8 Post-Second Vaccination: Missing | 0 | 1 | 1
  Day 22 Post-Second Vaccination: None | 20 | 19 | 19
  Day 22 Post-Second Vaccination: Mild (low) | 0 | 0 | 0
  Day 22 Post-Second Vaccination: Mild (high) | 1 | 0 | 0
  Day 22 Post-Second Vaccination: Moderate (low or high) | 0 | 0 | 0
  Day 22 Post-Second Vaccination: Severe (low or high) | 0 | 0 | 0
  Day 22 Post-Second Vaccination: Missing | 0 | 1 | 0
  Day 29 Post-Second Vaccination: None | 21 | 19 | 19
  Day 29 Post-Second Vaccination: Mild (low) | 0 | 0 | 0
  Day 29 Post-Second Vaccination: Mild (high) | 0 | 0 | 0
  Day 29 Post-Second Vaccination: Moderate (low or high) | 0 | 0 | 0
  Day 29 Post-Second Vaccination: Severe (low or high) | 0 | 0 | 0
  Day 29 Post-Second Vaccination: Missing | 0 | 1 | 0
  Max Severity Post Baseline: None | 20 | 20 | 19
  Max Severity Post Baseline: Mild (low) | 0 | 0 | 0
  Max Severity Post Baseline: Mild (high) | 1 | 0 | 0
  Max Severity Post Baseline: Moderate (low or high) | 0 | 0 | 0
  Max Severity Post Baseline: Severe (low or high) | 0 | 0 | 0
  Max Severity Post Baseline: Missing | 0 | 0 | 0

18. Primary Outcome: Number of Participants by Severity of Clinical Safety Laboratory Adverse Events - Potassium
Description: Thresholds for adverse events were considered as potassium 3.0 - 3.4 mmol/L or 5.2 - 6.0 mmol/L (mild), 2.5 - 2.9 mmol/L or 6.1 - 6.5 mmol/L (moderate), <2.5 mmol/L or >6.5 mmol/L (severe). If baseline clinical labs fell within mild range, then a laboratory AE was reported only if the value changed such that it fell into moderate range or higher when subsequent safety laboratory testing was done.
Time Frame: Day 1 to approximately 28 Days Post Second Vaccination
Population: Safety Population: includes all participants who received at least one study vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | ChAd3-EBO-Z + Placebo | ChAd3-EBO-Z + ChAd3-EBO-Z | ChAd3-EBO-Z + MVA- BN-Filo
Number analyzed (Participants) | 21 | 20 | 19
Participants
  Day 8 (Second Vaccination): None | 20 | 20 | 19
  Day 8 (Second Vaccination): Mild (low) | 0 | 0 | 0
  Day 8 (Second Vaccination): Mild (high) | 1 | 0 | 0
  Day 8 (Second Vaccination): Moderate (low or high) | 0 | 0 | 0
  Day 8 (Second Vaccination): Severe (low or high) | 0 | 0 | 0
  Day 8 (Second Vaccination): Missing | 0 | 0 | 0
  Day 8 Post-Second Vaccination: None | 20 | 19 | 18
  Day 8 Post-Second Vaccination: Mild (low) | 0 | 0 | 0
  Day 8 Post-Second Vaccination: Mild (high) | 1 | 0 | 0
  Day 8 Post-Second Vaccination: Moderate (low or high) | 0 | 0 | 0
  Day 8 Post-Second Vaccination: Severe (low or high) | 0 | 0 | 0
  Day 8 Post-Second Vaccination: Missing | 0 | 1 | 1
  Day 22 Post-Second Vaccination: None | 21 | 19 | 19
  Day 22 Post-Second Vaccination: Mild (low) | 0 | 0 | 0
  Day 22 Post-Second Vaccination: Mild (high) | 0 | 0 | 0
  Day 22 Post-Second Vaccination: Moderate (low or high) | 0 | 0 | 0
  Day 22 Post-Second Vaccination: Severe (low or high) | 0 | 0 | 0
  Day 22 Post-Second Vaccination: Missing | 0 | 1 | 0
  Day 29 Post-Second Vaccination: None | 20 | 19 | 19
  Day 29 Post-Second Vaccination: Mild (low) | 0 | 0 | 0
  Day 29 Post-Second Vaccination: Mild (high) | 1 | 0 | 0
  Day 29 Post-Second Vaccination: Moderate (low or high) | 0 | 0 | 0
  Day 29 Post-Second Vaccination: Severe (low or high) | 0 | 0 | 0
  Day 29 Post-Second Vaccination: Missing | 0 | 1 | 0
  Max Severity Post Baseline: None | 20 | 20 | 19
  Max Severity Post Baseline: Mild (low) | 0 | 0 | 0
  Max Severity Post Baseline: Mild (high) | 1 | 0 | 0
  Max Severity Post Baseline: Moderate (low or high) | 0 | 0 | 0
  Max Severity Post Baseline: Severe (low or high) | 0 | 0 | 0
  Max Severity Post Baseline: Missing | 0 | 0 | 0

19. Primary Outcome: Number of Participants by Severity of Clinical Safety Laboratory Adverse Events - BUN
Description: Thresholds for adverse events were considered as BUN 24 - 26 mg/dL (mild), 27 - 31 mg/dL (moderate), >31 mg/dL (severe). If baseline clinical labs fell within mild range, then a laboratory AE was reported only if the value changed such that it fell into moderate range or higher when subsequent safety laboratory testing was done.
Time Frame: Day 1 to approximately 28 Days Post Second Vaccination
Population: Safety Population: includes all participants who received at least one study vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | ChAd3-EBO-Z + Placebo | ChAd3-EBO-Z + ChAd3-EBO-Z | ChAd3-EBO-Z + MVA- BN-Filo
Number analyzed (Participants) | 21 | 20 | 19
Participants
  Day 8 (Second Vaccination): None | 1 | 3 | 1
  Day 8 (Second Vaccination): Mild | 0 | 0 | 0
  Day 8 (Second Vaccination): Moderate | 0 | 0 | 0
  Day 8 (Second Vaccination): Severe | 0 | 0 | 0
  Day 8 (Second Vaccination): Missing | 20 | 17 | 18
  Day 8 Post-Second Vaccination: None | 3 | 2 | 4
  Day 8 Post-Second Vaccination: Mild | 0 | 0 | 0
  Day 8 Post-Second Vaccination: Moderate | 0 | 0 | 0
  Day 8 Post-Second Vaccination: Severe | 0 | 0 | 0
  Day 8 Post-Second Vaccination: Missing | 18 | 18 | 15
  Day 22 Post-Second Vaccination: None | 2 | 2 | 0
  Day 22 Post-Second Vaccination: Mild | 0 | 0 | 0
  Day 22 Post-Second Vaccination: Moderate | 0 | 0 | 0
  Day 22 Post-Second Vaccination: Severe | 0 | 0 | 0
  Day 22 Post-Second Vaccination: Missing | 19 | 18 | 19
  Day 29 Post-Second Vaccination: None | 3 | 1 | 2
  Day 29 Post-Second Vaccination: Mild | 0 | 0 | 0
  Day 29 Post-Second Vaccination: Moderate | 0 | 0 | 0
  Day 29 Post-Second Vaccination: Severe | 0 | 0 | 0
  Day 29 Post-Second Vaccination: Missing | 18 | 19 | 17
  Max Severity Post Baseline: None | 4 | 3 | 4
  Max Severity Post Baseline: Mild | 0 | 0 | 0
  Max Severity Post Baseline: Moderate | 0 | 0 | 0
  Max Severity Post Baseline: Severe | 0 | 0 | 0
  Max Severity Post Baseline: Missing | 17 | 17 | 15

20. Primary Outcome: Number of Participants by Severity of Solicited Local Reactogenicity
Description: Local reactogenicity solicited on memory aid include pain; tenderness; pruritus (itch); erythema (redness), induration (hardness/swelling), and ecchymosis (bruising) (functional and measurement). Thresholds for severity were pain: aware, no interference with activity, no pain med (mild), aware, interferes with activity or requires repeated use of a non-narcotic pain reliever for >24 hr (moderate), aware, prevents activity or requires prescription med use (severe); tenderness: area surrounding injection hurts when touched or with arm motion, no interference with daily activity (mild), hurts when touched or with arm motion, interferes with activity (moderate), hurts when touched or with arm motion and prevents activity (severe); functional erythema, induration, ecchymosis, and pruritus: no activity interference (mild), interferes with activity (moderate), prevents activity (severe); erythema, induration, and ecchymosis (measurement): <20mm (mild), 20 - 50mm (moderate), >50mm (severe).
Time Frame: Day 1 to Day 8 Post First Vaccination
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | ChAd3-EBO-Z + Placebo | ChAd3-EBO-Z + ChAd3-EBO-Z | ChAd3-EBO-Z + MVABN-Filo
Number analyzed (Participants) | 21 | 20 | 19
Participants
  Any Local Symptom: None | 1 | 0 | 1
  Any Local Symptom: Mild | 17 | 17 | 11
  Any Local Symptom: Moderate | 3 | 2 | 5
  Any Local Symptom: Severe | 0 | 1 | 2
  Pain: None | 8 | 3 | 5
  Pain: Mild | 11 | 15 | 10
  Pain: Moderate | 2 | 2 | 3
  Pain: Severe | 0 | 0 | 1
  Tenderness: None | 4 | 1 | 4
  Tenderness: Mild | 16 | 18 | 12
  Tenderness: Moderate | 1 | 1 | 1
  Tenderness: Severe | 0 | 0 | 2
  Pruritus: None | 20 | 20 | 19
  Pruritus: Mild | 1 | 0 | 0
  Pruritus: Moderate | 0 | 0 | 0
  Pruritus: Severe | 0 | 0 | 0
  Ecchymosis (Functional grade): None | 21 | 18 | 17
  Ecchymosis (Functional grade): Mild | 0 | 2 | 2
  Ecchymosis (Functional grade): Moderate | 0 | 0 | 0
  Ecchymosis (Functional grade): Severe | 0 | 0 | 0
  Ecchymosis (Measurement grade): None | 21 | 18 | 17
  Ecchymosis (Measurement grade): Mild | 0 | 2 | 1
  Ecchymosis (Measurement grade): Moderate | 0 | 0 | 1
  Ecchymosis (Measurement grade): Severe | 0 | 0 | 0
  Erythema (Functional grade): None | 14 | 9 | 8
  Erythema (Functional grade): Mild | 7 | 10 | 11
  Erythema (Functional grade): Moderate | 0 | 1 | 0
  Erythema (Functional grade): Severe | 0 | 0 | 0
  Erythema (Measurement grade): None | 14 | 9 | 8
  Erythema (Measurement grade): Mild | 7 | 10 | 10
  Erythema (Measurement grade): Moderate | 0 | 0 | 1
  Erythema (Measurement grade): Severe | 0 | 1 | 0
  Induration (Functional grade): None | 15 | 13 | 14
  Induration (Functional grade): Mild | 6 | 6 | 3
  Induration (Functional grade): Moderate | 0 | 1 | 2
  Induration (Functional grade): Severe | 0 | 0 | 0
  Induration (Measurement grade): None | 15 | 13 | 14
  Induration (Measurement grade): Mild | 5 | 5 | 4
  Induration (Measurement grade): Moderate | 1 | 1 | 1
  Induration (Measurement grade): Severe | 0 | 1 | 0

21. Primary Outcome: Number of Participants by Severity of Solicited Local Reactogenicity
Description: Local reactogenicity solicited on memory aid include pain; tenderness; pruritus (itch); erythema (redness), induration (hardness/swelling), and ecchymosis (bruising) (functional and measurement). Thresholds for severity grading were pain: aware, no interference with activity, no pain med (mild), aware, interferes with activity or requires repeated use of a non-narcotic pain reliever for >24hr (moderate), aware, prevents activity or requires prescription med use (severe); tenderness: area surrounding injection hurts when touched or with arm motion, no interference with daily activity (mild), hurts when touched or with arm motion, interferes with activity (moderate), hurts when touched or with arm motion, prevents activity (severe); functional erythema, induration, ecchymosis, and pruritus: no activity interference (mild), interferes with activity (moderate), prevents activity (severe); erythema, induration, and ecchymosis (measurement): <20mm (mild), 20-50mm (moderate), >50mm (severe).
Time Frame: Day 1 to Day 8 Post Second Vaccination
Population: Safety Population Subset: includes all participants who received the first and second study vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | ChAd3-EBO-Z + Placebo | ChAd3-EBO-Z + ChAd3-EBO-Z | ChAd3-EBO-Z + MVA- BN-Filo
Number analyzed (Participants) | 17 | 17 | 18
Participants
  Any Local Symptom: None | 11 | 0 | 5
  Any Local Symptom: Mild | 6 | 10 | 13
  Any Local Symptom: Moderate | 0 | 6 | 0
  Any Local Symptom: Severe | 0 | 1 | 0
  Pain: None | 16 | 4 | 13
  Pain: Mild | 1 | 11 | 5
  Pain: Moderate | 0 | 2 | 0
  Pain: Severe | 0 | 0 | 0
  Tenderness: None | 14 | 2 | 6
  Tenderness: Mild | 3 | 9 | 12
  Tenderness: Moderate | 0 | 5 | 0
  Tenderness: Severe | 0 | 1 | 0
  Pruritus: None | 17 | 16 | 17
  Pruritus: Mild | 0 | 1 | 1
  Pruritus: Moderate | 0 | 0 | 0
  Pruritus: Severe | 0 | 0 | 0
  Ecchymosis (Functional grade): None | 17 | 17 | 18
  Ecchymosis (Functional grade): Mild | 0 | 0 | 0
  Ecchymosis (Functional grade): Moderate | 0 | 0 | 0
  Ecchymosis (Functional grade): Severe | 0 | 0 | 0
  Ecchymosis (Measurement grade): None | 17 | 17 | 18
  Ecchymosis (Measurement grade): Mild | 0 | 0 | 0
  Ecchymosis (Measurement grade): Moderate | 0 | 0 | 0
  Ecchymosis (Measurement grade): Severe | 0 | 0 | 0
  Erythema (Functional grade): None | 12 | 10 | 12
  Erythema (Functional grade): Mild | 5 | 7 | 6
  Erythema (Functional grade): Moderate | 0 | 0 | 0
  Erythema (Functional grade): Severe | 0 | 0 | 0
  Erythema (Measurement grade): None | 12 | 10 | 12
  Erythema (Measurement grade): Mild | 5 | 6 | 6
  Erythema (Measurement grade): Moderate | 0 | 1 | 0
  Erythema (Measurement grade): Severe | 0 | 0 | 0
  Induration (Functional grade): None | 17 | 14 | 17
  Induration (Functional grade): Mild | 0 | 3 | 1
  Induration (Functional grade): Moderate | 0 | 0 | 0
  Induration (Functional grade): Severe | 0 | 0 | 0
  Induration (Measurement grade): None | 17 | 14 | 17
  Induration (Measurement grade): Mild | 0 | 3 | 1
  Induration (Measurement grade): Moderate | 0 | 0 | 0
  Induration (Measurement grade): Severe | 0 | 0 | 0

22. Primary Outcome: Number of Participants by Severity of Solicited Local Reactogenicity
Description: as for outcome 21
Time Frame: Day 1 to Day 15
Population: Safety Population: includes all participants who received at least one study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | ChAd3-EBO-Z + Placebo | ChAd3-EBO-Z + ChAd3-EBO-Z | ChAd3-EBO-Z + MVA- BN-Filo
Number analyzed (Participants) | 21 | 20 | 19
Participants
  Any local symptom: Mild | 17 | 11 | 11
  Any local symptom: Moderate | 3 | 7 | 5
  Any local symptom: Severe | 0 | 2 | 2
  Any local symptom: None | 1 | 0 | 1
  Pain: Mild | 11 | 15 | 10
  Pain: Moderate | 2 | 3 | 3
  Pain: Severe | 0 | 0 | 1
  Pain: None | 8 | 2 | 5
  Tenderness: Mild | 16 | 12 | 12
  Tenderness: Moderate | 1 | 6 | 1
  Tenderness: Severe | 0 | 1 | 2
  Tenderness: None | 4 | 1 | 4
  Erythema (functional): Mild | 10 | 10 | 12
  Erythema (functional): Moderate | 0 | 1 | 0
  Erythema (functional): Severe | 0 | 0 | 0
  Erythema (functional): None | 11 | 9 | 7
  Erythema (measured): Mild | 10 | 9 | 11
  Erythema (measured): Moderate | 0 | 1 | 1
  Erythema (measured): Severe | 0 | 1 | 0
  Erythema (measured): None | 11 | 9 | 7
  Induration (functional): Mild | 6 | 7 | 3
  Induration (functional): Moderate | 0 | 1 | 2
  Induration (functional): Severe | 0 | 0 | 0
  Induration (functional): None | 15 | 12 | 14
  Induration (measured): Mild | 5 | 6 | 4
  Induration (measured): Moderate | 1 | 1 | 1
  Induration (measured): Severe | 0 | 1 | 0
  Induration (measured): None | 15 | 12 | 14
  Ecchymosis (functional): Mild | 0 | 2 | 2
  Ecchymosis (functional): Moderate | 0 | 0 | 0
  Ecchymosis (functional): Severe | 0 | 0 | 0
  Ecchymosis (functional): None | 21 | 18 | 17
  Ecchymosis (measured): Mild | 0 | 2 | 1
  Ecchymosis (measured): Moderate | 0 | 0 | 1
  Ecchymosis (measured): Severe | 0 | 0 | 0
  Ecchymosis (measured): None | 21 | 18 | 17
  Pruritus: Mild | 1 | 1 | 1
  Pruritus: Moderate | 0 | 0 | 0
  Pruritus: Severe | 0 | 0 | 0
  Pruritus: None | 20 | 19 | 18

23. Primary Outcome: Number of Participants by Severity of Solicited Systemic Reactogenicity
Description: Systemic reactogenicity solicited on memory aid included feverishness (chills/shivering/sweating), malaise (general unwell feeling), fatigue (tiredness), myalgia (body aches/muscular pain not at injection site), headache, nausea, loss of appetite, and elevated oral temperature. Thresholds for severity include feverishness, malaise, fatigue, myalgia, nausea, and loss of appetite: Noticeable but does not interfere with daily activity (Mild), Interferes with daily activity (Moderate), Significant interference, prevents daily activity (Severe); headache: Noticeable but does not interfere with daily activity (Mild), Any use of pain reliever or interferes with daily activity (Moderate), Significant interference, prevents daily activity, or requires any use of a prescription medication (Severe); elevated oral temperature: 37.8°C - 38.4°C or 100.00°F - 101.1°F (Mild), 38.5°C - 38.9°C or 101.2°F - 102.0°F (Moderate), >38.9°C or >102.0°F (Severe).
Time Frame: Day 1 to Day 8 Post First Vaccination
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | ChAd3-EBO-Z + Placebo | ChAd3-EBO-Z + ChAd3-EBO-Z | ChAd3-EBO-Z + MVABN-Filo
Number analyzed (Participants) | 21 | 20 | 19
Participants
  Any Systemic Symptom: None | 1 | 0 | 4
  Any Systemic Symptom: Mild | 7 | 8 | 3
  Any Systemic Symptom: Moderate | 7 | 5 | 6
  Any Systemic Symptom: Severe | 6 | 7 | 6
  Elevated Oral Temperature: None | 10 | 11 | 10
  Elevated Oral Temperature: Mild | 7 | 0 | 4
  Elevated Oral Temperature: Moderate | 2 | 3 | 3
  Elevated Oral Temperature: Severe | 2 | 6 | 2
  Feverishness: None | 6 | 6 | 6
  Feverishness: Mild | 5 | 6 | 5
  Feverishness: Moderate | 7 | 5 | 4
  Feverishness: Severe | 3 | 3 | 4
  Malaise: None | 8 | 3 | 6
  Malaise: Mild | 7 | 8 | 7
  Malaise: Moderate | 6 | 6 | 5
  Malaise: Severe | 0 | 3 | 1
  Fatigue: None | 4 | 5 | 6
  Fatigue: Mild | 13 | 6 | 7
  Fatigue: Moderate | 4 | 7 | 5
  Fatigue: Severe | 0 | 2 | 1
  Myalgia: None | 4 | 3 | 7
  Myalgia: Mild | 11 | 8 | 7
  Myalgia: Moderate | 6 | 7 | 4
  Myalgia: Severe | 0 | 2 | 1
  Headache: None | 11 | 10 | 7
  Headache: Mild | 9 | 3 | 8
  Headache: Moderate | 1 | 6 | 4
  Headache: Severe | 0 | 1 | 0
  Nausea: None | 15 | 11 | 16
  Nausea: Mild | 5 | 7 | 2
  Nausea: Moderate | 0 | 2 | 1
  Nausea: Severe | 1 | 0 | 0
  Loss of Appetite: None | 17 | 11 | 11
  Loss of Appetite: Mild | 2 | 8 | 5
  Loss of Appetite: Moderate | 2 | 1 | 3
  Loss of Appetite: Severe | 0 | 0 | 0

24. Primary Outcome: Number of Participants by Severity of Solicited Systemic Reactogenicity
Description: as for outcome 23
Time Frame: Day 1 to Day 8 Post Second Vaccination
Population: Safety Population Subset: includes all participants who received the first and second study vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | ChAd3-EBO-Z + Placebo | ChAd3-EBO-Z + ChAd3-EBO-Z | ChAd3-EBO-Z + MVA- BN-Filo
Number analyzed (Participants) | 17 | 17 | 18
Participants
  Any Systemic Symptom: None | 9 | 3 | 12
  Any Systemic Symptom: Mild | 6 | 5 | 4
  Any Systemic Symptom: Moderate | 2 | 6 | 2
  Any Systemic Symptom: Severe | 0 | 3 | 0
  Elevated Oral Temperature: None | 17 | 9 | 18
  Elevated Oral Temperature: Mild | 0 | 6 | 0
  Elevated Oral Temperature: Moderate | 0 | 1 | 0
  Elevated Oral Temperature: Severe | 0 | 1 | 0
  Feverishness: None | 14 | 6 | 17
  Feverishness: Mild | 2 | 7 | 1
  Feverishness: Moderate | 1 | 3 | 0
  Feverishness: Severe | 0 | 1 | 0
  Malaise: None | 14 | 3 | 17
  Malaise: Mild | 2 | 9 | 1
  Malaise: Moderate | 1 | 4 | 0
  Malaise: Severe | 0 | 1 | 0
  Fatigue: None | 10 | 3 | 15
  Fatigue: Mild | 6 | 9 | 2
  Fatigue: Moderate | 1 | 4 | 1
  Fatigue: Severe | 0 | 1 | 0
  Myalgia: None | 14 | 6 | 14
  Myalgia: Mild | 2 | 4 | 4
  Myalgia: Moderate | 1 | 6 | 0
  Myalgia: Severe | 0 | 1 | 0
  Headache: None | 10 | 8 | 14
  Headache: Mild | 6 | 6 | 3
  Headache: Moderate | 1 | 3 | 1
  Headache: Severe | 0 | 0 | 0
  Nausea: None | 15 | 13 | 17
  Nausea: Mild | 2 | 3 | 0
  Nausea: Moderate | 0 | 1 | 1
  Nausea: Severe | 0 | 0 | 0
  Loss of Appetite: None | 14 | 10 | 18
  Loss of Appetite: Mild | 3 | 7 | 0
  Loss of Appetite: Moderate | 0 | 0 | 0
  Loss of Appetite: Severe | 0 | 0 | 0

25. Primary Outcome: Number of Participants by Severity of Solicited Systemic Reactogenicity
Description: as for outcome 23
Time Frame: Day 1 to Day 15
Population: Safety Population: includes all participants who received at least one study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | ChAd3-EBO-Z + Placebo | ChAd3-EBO-Z + ChAd3-EBO-Z | ChAd3-EBO-Z + MVA- BN-Filo
Number analyzed (Participants) | 21 | 20 | 19
Participants
  Any Systemic Symptom: Mild | 6 | 6 | 3
  Any Systemic Symptom: Moderate | 8 | 7 | 6
  Any Systemic Symptom: Severe | 6 | 7 | 6
  Any Systemic Symptom: None | 1 | 0 | 4
  Elevated Oral Temperature: Mild | 7 | 3 | 4
  Elevated Oral Temperature: Moderate | 2 | 3 | 3
  Elevated Oral Temperature: Severe | 2 | 6 | 2
  Elevated Oral Temperature: None | 10 | 8 | 10
  Feverishness: Mild | 7 | 7 | 5
  Feverishness: Moderate | 8 | 6 | 4
  Feverishness: Severe | 3 | 3 | 4
  Feverishness: None | 3 | 4 | 6
  Malaise: Mild | 7 | 10 | 7
  Malaise: Moderate | 7 | 5 | 5
  Malaise: Severe | 0 | 4 | 1
  Malaise: None | 7 | 1 | 6
  Fatigue: Mild | 13 | 9 | 7
  Fatigue: Moderate | 5 | 8 | 5
  Fatigue: Severe | 0 | 2 | 1
  Fatigue: None | 3 | 1 | 6
  Myalgia: Mild | 10 | 8 | 7
  Myalgia: Moderate | 7 | 9 | 4
  Myalgia: Severe | 0 | 3 | 1
  Myalgia: None | 4 | 0 | 7
  Headache: Mild | 11 | 5 | 8
  Headache: Moderate | 2 | 7 | 4
  Headache: Severe | 0 | 1 | 0
  Headache: None | 8 | 7 | 7
  Nausea: Mild | 6 | 7 | 1
  Nausea: Moderate | 0 | 3 | 2
  Nausea: Severe | 1 | 0 | 0
  Nausea: None | 14 | 10 | 16
  Loss of Appetite: Mild | 4 | 11 | 5
  Loss of Appetite: Moderate | 2 | 1 | 3
  Loss of Appetite: Severe | 0 | 0 | 0
  Loss of Appetite: None | 15 | 8 | 11

26. Primary Outcome: Number of Participants by Severity of Vaccine-related Unsolicited Adverse Events (AEs)
Description: Vaccine-related unsolicited AEs include any untoward medical occurrence in a participant for which there is evidence to suggest a causal relationship between the study product and the adverse event. Thresholds for severity include events require minimal or no treatment and do not interfere with the subject's daily activities (mild), events result in a low level of inconvenience or concern with therapeutic measures and may cause some interference with functioning and daily activities (moderate), and events interrupt the subject's daily activities and may require systemic drug therapy or other treatment and are usually incapacitating (severe). Participants are counted once per preferred term and are summarized according to their highest severity. No severe events were reported.
Time Frame: Day 1 to approximately 28 Days Post Second Vaccination
Population: Safety Population: includes all participants who received at least one study vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | ChAd3-EBO-Z + Placebo | ChAd3-EBO-Z + ChAd3-EBO-Z | ChAd3-EBO-Z + MVA- BN-Filo
Number analyzed (Participants) | 21 | 20 | 19
Participants
  Any Event: Mild | 3 | 7 | 4
  Any Event: Moderate | 1 | 3 | 0
  Any Event: None | 17 | 10 | 15
  Lymphadenopathy: Mild | 0 | 1 | 1
  Lymphadenopathy: Moderate | 1 | 0 | 0
  Lymphadenopathy: None | 20 | 19 | 18
  Tachycardia: Mild | 0 | 1 | 0
  Tachycardia: Moderate | 0 | 0 | 0
  Tachycardia: None | 21 | 19 | 19
  Diarrhea: Mild | 0 | 0 | 0
  Diarrhea: Moderate | 0 | 1 | 0
  Diarrhea: None | 21 | 19 | 19
  Vomiting: Mild | 1 | 1 | 1
  Vomiting: Moderate | 0 | 1 | 0
  Vomiting: None | 20 | 18 | 18
  Chest discomfort: Mild | 0 | 0 | 0
  Chest discomfort: Moderate | 0 | 1 | 0
  Chest discomfort: None | 21 | 19 | 19
  Blood pressure diastolic decreased: Mild | 0 | 0 | 1
  Blood pressure diastolic decreased: Moderate | 0 | 0 | 0
  Blood pressure diastolic decreased: None | 21 | 20 | 18
  Transaminases increased: Mild | 0 | 0 | 0
  Transaminases increased: Moderate | 0 | 1 | 0
  Transaminases increased: None | 21 | 19 | 19
  Dehydration: Mild | 0 | 1 | 0
  Dehydration: Moderate | 0 | 0 | 0
  Dehydration: None | 21 | 19 | 19
  Back pain: Mild | 0 | 1 | 0
  Back pain: Moderate | 0 | 0 | 0
  Back pain: None | 21 | 19 | 19
  Muscle Spasms: Mild | 0 | 0 | 1
  Muscle Spasms: Moderate | 0 | 0 | 0
  Muscle Spasms: None | 21 | 20 | 18
  Dizziness: Mild | 0 | 1 | 0
  Dizziness: Moderate | 0 | 0 | 0
  Dizziness: None | 21 | 19 | 19
  Sinus headache: Mild | 1 | 0 | 0
  Sinus headache: Moderate | 0 | 0 | 0
  Sinus headache: None | 20 | 20 | 19
  Taste Disorder: Mild | 0 | 1 | 0
  Taste Disorder: Moderate | 0 | 0 | 0
  Taste Disorder: None | 21 | 19 | 19
  Cough: Mild | 1 | 0 | 0
  Cough: Moderate | 0 | 0 | 0
  Cough: None | 20 | 20 | 19
  Oropharyngeal pain: Mild | 1 | 0 | 0
  Oropharyngeal pain: Moderate | 0 | 0 | 0
  Oropharyngeal pain: None | 20 | 20 | 19
  Sinus Congestion: Mild | 0 | 1 | 0
  Sinus Congestion: Moderate | 0 | 0 | 0
  Sinus Congestion: None | 21 | 19 | 19
  Acne: Mild | 0 | 1 | 0
  Acne: Moderate | 0 | 0 | 0
  Acne: None | 21 | 19 | 19
  Ecchymosis: Mild | 0 | 1 | 0
  Ecchymosis: Moderate | 0 | 0 | 0
  Ecchymosis: None | 21 | 19 | 19
  Rash: Mild | 0 | 1 | 0
  Rash: Moderate | 0 | 0 | 0
  Rash: None | 21 | 19 | 19

27. Secondary Outcome: Geometric Mean Fold Rise (GMFR) as Measured by Anti-EBOV GP ELISA - ITT Population
Description: The endpoint assessed antibodies against Ebola virus (EBOV) glycoproteins (GP) using an enzyme-linked immunosorbent assay (anti-EBOV GP ELISA). Venous blood samples for serum were used for this assay. Geometric mean fold rise (GMFR) compared to baseline (Day 1) was calculated for each study arm.
Time Frame: Day 8, 15, 22, 29 and 36 compared to baseline (Day 1) reported as Day 8 post-first vaccination, Day 8 post-second vaccination, Day 15 post-second vaccination, Day 22 post-second vaccination, and Day 29 post-second vaccination, respectively.
Population: ITT Population: includes all participants who received at least one study vaccination and contributed both pre- and at least one post-study vaccination blood samples for immunogenicity testing for which valid results were reported
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | ChAd3-EBO-Z + Placebo | ChAd3-EBO-Z + ChAd3-EBO-Z | ChAd3-EBO-Z + MVA- BN-Filo
Number analyzed (Participants) | 21 | 19 | 19
titer
  Day 8 Post-First Vaccination (Second Vaccination): number analyzed (Participants) | 21 | 19 | 18
  Day 8 Post-First Vaccination (Second Vaccination) | 1.1 [0.9 to 1.3] | 1.2 [0.8 to 1.7] | 1.3 [0.8 to 1.9]
  Day 8 Post-Second Vaccination: number analyzed (Participants) | 21 | 18 | 18
  Day 8 Post-Second Vaccination | 21.5 [13.3 to 35.0] | 21.0 [11.9 to 37.0] | 25.4 [11.3 to 57.1]
  Day 15 Post-Second Vaccination: number analyzed (Participants) | 21 | 18 | 19
  Day 15 Post-Second Vaccination | 54.3 [32.3 to 91.0] | 54.9 [28.2 to 106.6] | 49.6 [25.6 to 96.0]
  Day 22 Post-Second Vaccination: number analyzed (Participants) | 21 | 18 | 19
  Day 22 Post-Second Vaccination | 70.7 [41.2 to 121.2] | 77.6 [40.3 to 149.5] | 74.1 [37.4 to 146.6]
  Day 29 Post-Second Vaccination: number analyzed (Participants) | 21 | 18 | 19
  Day 29 Post-Second Vaccination | 83.3 [44.9 to 154.8] | 97.8 [52.2 to 183.0] | 82.6 [38.8 to 176.1]

28. Secondary Outcome: Geometric Mean Fold Rise (GMFR) as Measured by Anti-EBOV GP ELISA - Per Prototocol Population
Description: as for outcome 27
Time Frame: as for outcome 27
Population: Per Protocol population includes all participants who received at least one study vaccination, contributed both pre- and at least one post-study vaccination blood samples for immunogenicity testing for which valid results were reported, were eligible at baseline and have no major protocol deviations.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | ChAd3-EBO-Z + Placebo | ChAd3-EBO-Z + ChAd3-EBO-Z | ChAd3-EBO-Z + MVA- BN-Filo
Number analyzed (Participants) | 21 | 19 | 19
titer
  Day 8 Post-First Vaccination (Second Vaccination): number analyzed (Participants) | 21 | 19 | 18
  Day 8 Post-First Vaccination (Second Vaccination) | 1.1 [0.9 to 1.3] | 1.2 [0.8 to 1.7] | 1.3 [0.8 to 1.9]
  Day 8 Post-Second Vaccination: number analyzed (Participants) | 17 | 16 | 17
  Day 8 Post-Second Vaccination | 25.1 [15.2 to 41.4] | 17.4 [9.9 to 30.9] | 23.1 [10.0 to 53.3]
  Day 15 Post-Second Vaccination: number analyzed (Participants) | 16 | 16 | 18
  Day 15 Post-Second Vaccination | 61.3 [33.3 to 112.8] | 45.3 [24.0 to 85.2] | 43.5 [23.0 to 82.5]
  Day 22 Post-Second Vaccination: number analyzed (Participants) | 17 | 16 | 17
  Day 22 Post-Second Vaccination | 75.3 [42.0 to 135.2] | 66.8 [33.4 to 133.8] | 64.0 [32.1 to 127.6]
  Day 29 Post-Second Vaccination: number analyzed (Participants) | 17 | 16 | 17
  Day 29 Post-Second Vaccination | 92.4 [46.3 to 184.4] | 83.0 [44.2 to 156.0] | 66.7 [30.8 to 144.2]

29. Secondary Outcome: Geometric Mean Titer (GMT) as Measured by Anti-EBOV GP ELISA - ITT Population
Description: The endpoint assessed antibodies against Ebola virus (EBOV) glycoproteins (GP) using an enzyme-linked immunosorbent assay (anti-EBOV GP ELISA). Venous blood samples for serum were used for this assay. Geometric Mean Titer (GMT) was calculated for each study arm.
Time Frame: Day 1, 8, 15, 22, 29 and 36 reported as Day 1 first vaccination, Day 8 post-first vaccination, Day 8 post-second vaccination, Day 15 post-second vaccination, Day 22 post-second vaccination, and Day 29 post-second vaccination, respectively.
Population: as for outcome 27
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | ChAd3-EBO-Z + Placebo | ChAd3-EBO-Z + ChAd3-EBO-Z | ChAd3-EBO-Z + MVA- BN-Filo
Number analyzed (Participants) | 21 | 19 | 19
titer
  Day 1 First Vaccination | 29.5 [23.1 to 37.6] | 33.5 [23.0 to 48.7] | 32.3 [23.0 to 45.3]
  Day 8 Post-First Vaccination (Second Vaccination): number analyzed (Participants) | 21 | 19 | 18
  Day 8 Post-First Vaccination (Second Vaccination) | 32.6 [23.9 to 44.3] | 40.2 [26.9 to 60.1] | 35.4 [23.0 to 54.4]
  Day 8 Post-Second Vaccination: number analyzed (Participants) | 21 | 18 | 18
  Day 8 Post-Second Vaccination | 635.0 [424.3 to 950.3] | 712.7 [413.3 to 1229.2] | 831.4 [411.2 to 1681.2]
  Day 15 Post-Second Vaccination: number analyzed (Participants) | 21 | 18 | 19
  Day 15 Post-Second Vaccination | 1600.0 [1012.9 to 2527.5] | 1866.4 [1003.4 to 3471.8] | 1600.0 [937.9 to 2729.4]
  Day 22 Post-Second Vaccination: number analyzed (Participants) | 21 | 18 | 19
  Day 22 Post-Second Vaccination | 2083.5 [1312.2 to 3308.3] | 2639.6 [1539.3 to 4526.2] | 2390.0 [1483.9 to 3849.3]
  Day 29 Post-Second Vaccination: number analyzed (Participants) | 21 | 18 | 19
  Day 29 Post-Second Vaccination | 2457.4 [1456.6 to 4145.8] | 3325.6 [1898.7 to 5824.8] | 2666.4 [1497.5 to 4747.9]

30. Secondary Outcome: Geometric Mean Titer (GMT) as Measured by Anti-EBOV GP ELISA - Per Protocol Population
Description: as for outcome 29
Time Frame: as for outcome 29
Population: as for outcome 28
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | ChAd3-EBO-Z + Placebo | ChAd3-EBO-Z + ChAd3-EBO-Z | ChAd3-EBO-Z + MVA- BN-Filo
Number analyzed (Participants) | 21 | 19 | 19
titer
  Day 1 First Vaccination | 29.5 [23.1 to 37.6] | 33.5 [23.0 to 48.7] | 32.3 [23.0 to 45.3]
  Day 8 Post-First Vaccination (Second Vaccination): number analyzed (Participants) | 21 | 19 | 18
  Day 8 Post-First Vaccination (Second Vaccination) | 32.6 [23.9 to 44.3] | 40.2 [26.9 to 60.1] | 35.4 [23.0 to 54.4]
  Day 8 Post-Second Vaccination: number analyzed (Participants) | 17 | 16 | 17
  Day 8 Post-Second Vaccination | 679.6 [420.4 to 1098.6] | 590.7 [344.6 to 1012.6] | 768.0 [370.5 to 1592.1]
  Day 15 Post-Second Vaccination: number analyzed (Participants) | 16 | 16 | 18
  Day 15 Post-Second Vaccination | 1670.8 [935.9 to 2983.0] | 1532.2 [845.0 to 2778.1] | 1425.4 [860.2 to 2362.1]
  Day 22 Post-Second Vaccination: number analyzed (Participants) | 17 | 16 | 17
  Day 22 Post-Second Vaccination | 2043.5 [1180.9 to 3536.1] | 2262.7 [1297.6 to 3945.8] | 2128.5 [1374.2 to 3296.8]
  Day 29 Post-Second Vaccination: number analyzed (Participants) | 17 | 16 | 17
  Day 29 Post-Second Vaccination | 2505.6 [1335.4 to 4701.0] | 2810.0 [1605.7 to 4917.6] | 2217.1 [1259.9 to 3901.4]

31. Secondary Outcome: Seroconversion as Measured by Anti-EBOV GP ELISA - ITT Population
Description: The endpoint assessed antibodies against Ebola virus (EBOV) glycoproteins (GP) using an enzyme-linked immunosorbent assay (anti-EBOV GP ELISA). Venous blood samples for serum were used for this assay. Seroconversion was calculated for each study arm and was defined as anti-EBOV GP ELISA titer > 50 if baseline (Day 1) titer = 50 or fold rise > 4 as compared to baseline if baseline titer > 50.
Time Frame: Day 8, 15, 22, 29 and 36 reported as Day 8 post-first vaccination, Day 8 post-second vaccination, Day 15 post-second vaccination, Day 22 post-second vaccination, and Day 29 post-second vaccination, respectively.
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | ChAd3-EBO-Z + Placebo | ChAd3-EBO-Z + ChAd3-EBO-Z | ChAd3-EBO-Z + MVA- BN-Filo
Number analyzed (Participants) | 21 | 19 | 19
Participants
  Day 8 Post-First Vaccination (Second Vaccination): number analyzed (Participants) | 21 | 19 | 18
  Day 8 Post-First Vaccination (Second Vaccination) | 1 | 2 | 1
  Day 8 Post-Second Vaccination: number analyzed (Participants) | 21 | 18 | 18
  Day 8 Post-Second Vaccination | 20 | 17 | 17
  Day 15 Post-Second Vaccination: number analyzed (Participants) | 21 | 18 | 19
  Day 15 Post-Second Vaccination | 21 | 17 | 19
  Day 22 Post-Second Vaccination: number analyzed (Participants) | 21 | 18 | 19
  Day 22 Post-Second Vaccination | 21 | 17 | 18
  Day 29 Post-Second Vaccination: number analyzed (Participants) | 21 | 18 | 19
  Day 29 Post-Second Vaccination | 21 | 18 | 18

32. Secondary Outcome: Seroconversion as Measured by Anti-EBOV GP ELISA - Per Protocol Population
Description: as for outcome 31
Time Frame: as for outcome 31
Population: as for outcome 28
Measure: Count of Participants; unit: Participants
Arm/Group | ChAd3-EBO-Z + Placebo | ChAd3-EBO-Z + ChAd3-EBO-Z | ChAd3-EBO-Z + MVA- BN-Filo
Number analyzed (Participants) | 21 | 19 | 19
Participants
  Day 8 Post-First Vaccination (Second Vaccination): number analyzed (Participants) | 21 | 19 | 18
  Day 8 Post-First Vaccination (Second Vaccination) | 1 | 2 | 1
  Day 8 Post-Second Vaccination: number analyzed (Participants) | 17 | 16 | 17
  Day 8 Post-Second Vaccination | 17 | 15 | 16
  Day 15 Post-Second Vaccination: number analyzed (Participants) | 16 | 16 | 18
  Day 15 Post-Second Vaccination | 16 | 15 | 18
  Day 22 Post-Second Vaccination: number analyzed (Participants) | 17 | 16 | 17
  Day 22 Post-Second Vaccination | 17 | 15 | 16
  Day 29 Post-Second Vaccination: number analyzed (Participants) | 17 | 16 | 17
  Day 29 Post-Second Vaccination | 17 | 16 | 16

ADVERSE EVENTS:
Time Frame: Solicited events were collected from the time of each study vaccination through 7 days post-vaccination. Vaccine-related unsolicited events were collected from the first study vaccination through 28 days post second vaccination. Clinical safety laboratory events were collected from the time of first study vaccination through approximately 28 days after the second vaccination. SAEs and vaccine-related MAAEs were collected through 6 months post the first vaccination.
Description: The solicited and unsolicited adverse events were assessed using MedDRA 23.0.
Arm/Group | ChAd3-EBO-Z + Placebo | ChAd3-EBO-Z + ChAd3-EBO-Z | ChAd3-EBO-Z + MVA- BN-Filo
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/20 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 21/21 | 20/20 | 19/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ChAd3-EBO-Z + Placebo (N=21) | ChAd3-EBO-Z + ChAd3-EBO-Z (N=20) | ChAd3-EBO-Z + MVA- BN-Filo (N=19)
Pyrexia (General disorders) | 11 (11) | 12 (17) | 9 (9)
Malaise (General disorders) | 14 (16) | 19 (31) | 13 (14)
Fatigue (General disorders) | 18 (24) | 19 (29) | 13 (16)
Myalgia (Musculoskeletal and connective tissue disorders) | 17 (20) | 20 (28) | 12 (16)
Headache (General disorders) | 13 (17) | 13 (19) | 12 (16)
Nausea (General disorders) | 7 (8) | 10 (13) | 3 (4)
Decreased Appetite (Metabolism and nutrition disorders) | 6 (7) | 12 (16) | 8 (8)
Vulvovaginal Pruritus (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Blood Pressure Diastolic Decreased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Chest Discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Feeling Of Body Temperature Change (General disorders) | 18 (18) | 16 (25) | 13 (14)
Injection Site Haemorrhage (General disorders) | 0 (0) | 2 (2) | 2 (2)
Ligament Rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Limb Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (3) | 1 (1) | 1 (1)
Muscle Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Taste Disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Tibia Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Transaminases Increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 1 (1) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Vaccination Site Erythema (General disorders) | 10 (12) | 11 (18) | 12 (17)
Vaccination Site Induration (General disorders) | 6 (6) | 8 (10) | 5 (6)
Vaccination Site Pain (General disorders) | 18 (21) | 20 (37) | 18 (31)
Vaccination Site Pruritus (General disorders) | 1 (1) | 1 (1) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 1 (2) | 2 (2) | 1 (1)
Blood Creatinine Increased (Investigations) | 2 (2) | 1 (1) | 2 (2)
Haemoglobin Decreased (Investigations) | 2 (4) | 6 (6) | 2 (3)
Neutrophil Count Decreased (Investigations) | 1 (1) | 5 (6) | 3 (4)
Platelet Count Decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
White Blood Cell Count Decreased (Investigations) | 2 (4) | 4 (5) | 4 (5)
White Blood Cell Count Increased (Investigations) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-01-30): https://cdn.clinicaltrials.gov/large-docs/06/NCT03583606/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-29): https://cdn.clinicaltrials.gov/large-docs/06/NCT03583606/SAP_001.pdf